CLINICAL TRIAL: NCT04761692
Title: Improving Vaccine Acceptance and Uptake Among Underresourced African American and Latinx Older Adults: A Multidisciplinary and Culturally Based Training Program for Minority Churches
Brief Title: Increasing COVID-19, Influenza, and Pneumonia Vaccine Uptake
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: vaccineinc
Record Dates: First submitted 2021-02-02; First posted 2021-02-21 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Covid19; Influenza; Pneumonia; Vaccine Refusal
Keywords: African American; Latinx; Vaccine; Hispanic; Latino; COVID19 Vaccine
MeSH Terms: conditions — COVID-19; Influenza, Human; Pneumonia; Vaccination Refusal

STUDY DESIGN:
Intervention Model Description: The VEPMP will consist of recruited churches in 15 cohorts of 2 churches per cohort (total n = 30). Each cohort of church will include an AA and a Latinx church. The 15 church cohorts will be randomized to three arms based on a 1:1:1 ratio, using an online random number generator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): This arm will include 5 churches who will receive all study activities in the Vaccine Education Promotion Management Plan
  Interventions: Behavioral: Full VEPMP Intervention
- Arm 2 (Experimental): This arm will include 5 churches who will receive some study activities in the Vaccine Education Promotion Management Plan
  Interventions: Behavioral: Partial VEPMP Intervention
- Arm 3 (Experimental): This arm will include 5 churches who will receive all study activities in the Vaccine Education Promotion Management Plan following completion of Arm 1 and 2.
  Interventions: Behavioral: Delayed VEPMP Intervention

INTERVENTIONS:
Behavioral: Full VEPMP Intervention — Delivery of intrapersonal/interpersonal (i.e., motivational interviewing, vaccine educators, personal testimony, etc.), AND organizational (i.e., church-based sponsored events, seminars, web/online activities, bulletin inserts, etc.)
  Arms: Arm 1
Behavioral: Partial VEPMP Intervention — Delivery of iAND organizational (i.e., church-based sponsored events, seminars, web/online activities, bulletin inserts, etc.)
  Arms: Arm 2
Behavioral: Delayed VEPMP Intervention — Delayed implementation of delivery of intrapersonal/interpersonal AND organizational after 1 year of study start
  Arms: Arm 3

SUMMARY:
This proposed study seeks to community knowledge and understand the experience of underserved communities in the exploration of reducing health disparities and increasing vaccine uptake and acceptability COVID-19, influenza, and pneumonia for AA and Latinx populations. Unique in its design, it has the following characteristics: 1) multifaceted, 2) culturally tailored, 3) community-based, and 4) mixed methods in which the outcomes of interest will be measured before and after the intervention with 18-month interval. Furthermore, we seek to enhance our partnerships and collaborations with churches in South Los Angeles by supporting efforts to encourage COVID-19, influenza, and pneumonia vaccination uptake among underserved minorities in one of the most challenged and hard-to-reach population areas in the nation.

DETAILED DESCRIPTION:
This study seeks to augment community knowledge and increase vaccine uptake among under-resourced African American and Latinx communities in South LA via leveraging trusted church leaders, educators and influencers to delivering COVID-19, influenza, and pneumonia education on vaccination. Unique in its design, this study has the following characteristics, beneficial to the acceptability and success of the proposal, it is: 1) multifaceted, 2) culturally tailored, and 3) community-based, in which the outcomes of interest will be compared longitudinally between arms 1-3, including measurement before and after the intervention with 9- and 18-month interval.

ELIGIBILITY:
Inclusion Criteria:

* Parishioner at a church receiving the VEPMP intervention
* Identify as African American or Latinx,
* at least 65 years and older
* Have Not received a vaccine for COVID-19, influenza, or pneumonia within the previous 24 months
* Agrees to study terms, which include follow-up interviews 9 and 18 months after study enrollment

Exclusion Criteria:

* Does not attend or identify as a Parishioner at a church receiving the VEPMP intervention
* Does not identify as African American or Latinx
* Under the age of 65 years
* Received all vaccine doses for COVID-19, influenza, or pneumonia within the previous 24 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of vaccination uptake for COVID-19, influenza, and pneumonia using Vaccination History Self Report | Intervention: 12 months; Follow-up Point: 9 & 18 months post-intervention
  By comparison of pre-, post- intervention, and 9- and 18-months follow-up data, we anticipate the following compared to baseline: a 30% change in uptake for vaccination.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Adherence to COVID-19, influenza, and pneumonia vaccination schedules Risk Using the NIH Toolbox Surveys on COVID-19 | Intervention: 12 months; Follow-up Point: 9 & 18 months post-intervention
  By comparison of pre-, post- intervention, and 9 and 18-months follow-up data, we anticipate the following compared to baseline: a 30% change in adherence to COVID-19, influenza, and pneumonia vaccination schedules.
Percentage of Participants Achieving Decreased Vaccine Hesitancy Levels of COVID-19, influenza, and pneumonia Using the NIH Toolbox Surveys on COVID-19, influenza, and pneumonia | Intervention: 12 months; Follow-up Point: 9 & 18 months post-intervention
  By comparison of pre-, post- intervention, and 9 and 18-months follow-up data, we anticipate the following compared to baseline: a 40% change in vaccine hesitancy toward COVID-19, influenza, and pneumonia vaccination
Percentage of Participants Achieving Decreased Levels of COVID-19, influenza, and pneumonia Mistrust and Barriers Using the NIH Toolbox Surveys on COVID-19, influenza, and pneumonia | Intervention: 12 months; Follow-up Point: 9 & 18 months post-intervention
  By comparison of pre-, post- intervention, and 9 and 18-months follow-up data, we anticipate the following compared to baseline: a 40% change in mistrust and perceived barriers toward COVID-19, influenza, and pneumonia vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Bazargan, PhD, Principal Investigator — Charles R. Drew University of Medicine & Science
Locations (1):
- Charles R. Drew University of Medicine & Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No